CLINICAL TRIAL: NCT05303948
Title: Evaluation and Comparison of Two Positions for Free Floating Tracheal Intubation in Weightlessness: An Ice-Pick Position With a Direct Laryngoscopy and the Classic Approach With VideolaryngoscopyY
Brief Title: Evaluation of Two Positions for Free Floating Tracheal Intubation in Weightlessness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier de Bretagne Sud (Other)
Collaborators: Centre National d'Etudes Spatiales (Other Government)
Responsible Party: Principal Investigator, Dr Seamus Thierry, Anesthesiologist and Intensive Care Doctor, Groupe Hospitalier de Bretagne Sud
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2019-1
Record Dates: First submitted 2022-02-22; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Intubation; Difficult or Failed; Intubation Complication

STUDY DESIGN:
Intervention Model Description: A simulation study, in which participants alternatively perform oro-tracheal intubation on a manikin, either using a videolaryngoscope (McGrath model, Medtronic TM) or a direct laryngoscope
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct laryngoscopy in the ice-pick position (Experimental): In this arm, participants are assigned to intubations attempts in weightlessness on a manikin.
  The insertion of a 7.0 mm cuffed oro-tracheal tube was performed by using a direct laryngoscope with a Macintosh non-angulated size 3 blade, in a "face-to-face" or ice-pick position.
  Interventions: Device: Videolaryngoscopy / Direct Laryngoscopy
- Video-laryngoscopy in free-floating position (Experimental): In this arm, participants are assigned to intubations attempts in weightlessness on a manikin.
  The insertion of a 7.0 mm cuffed oro-tracheal tube was performed by using a video laryngoscopy in a semi-free-floating position (McGrath model, Covidien™, Medtronic™).
  Interventions: Device: Videolaryngoscopy / Direct Laryngoscopy

INTERVENTIONS:
Device: Videolaryngoscopy / Direct Laryngoscopy — First pass success analysis

SUMMARY:
In a non-randomized, controlled, cross-over simulation study, the investigators evaluated and compared intubation performance of trained operators, using either a conventional laryngoscope in an ice-pick position or a video laryngoscope in a free-floating classic position, in weightlessness and in normogravity.

Data were analyzed with the generalized linear mixed-effects models.

Primary endpoint was the success rate of tracheal intubation. Time to intubation and the confidence score into the success of tube placement were also recorded as secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers

* aged between 18 and 65 years old.
* Absence of pregnancy
* Belonging to a Health Insurance Coverage by the French Social Security Program or equivalent, proved by a European Health Insurance Card (EHIC).
* Medically fit to fly after a JAR FCL3 - Class 2 examination

Exclusion Criteria before the flight

* positive pregnancy test on flight day
* anxiety
* non-participation in flight safety briefing

Exclusion Criteria during the flight

* failure to follow safety guidelines
* occurence of motion sickness during the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-10-18 (Actual)

PRIMARY OUTCOMES:
First pass success | 1 day (1 flight)
  Bi-pulmonary ventilation success was assessed by the intubating operator performing chest auscultation and by the measurement of a tidal volume on the mannequin's electronic sensors. Selective side intubation was considered as failure

SECONDARY OUTCOMES:
Time | 1 day (1 flight)
  The duration (seconds) of each attempt was recorded and ended with vocal confirmation of tube placement from the intubating operator or at the end of the parabola
Confidence Score | 1 day (1 flight)
  A subjective score of confidence in the correct tube placement was recorded after each attempt and ranked from minus ten (complete certainty about failure) to plus ten (complete certainty about success). A score of zero was pronounced by the operator when he/she had maximum uncertainty about success or failure.

CONTACTS AND LOCATIONS:
Overall Officials: Séamus Thierry, MD, Principal Investigator — Groupe Hospitalier de Bretagne Sud
Locations (1):
- Groupe Hospitalier de Bretagne Sud, Lorient, France

IPD SHARING:
Plan to Share IPD: Yes
All relevant data, anonymized, will be available from Dr S.Thierry on request
Supporting Information: Study Protocol, SAP, Analytic Code

REFERENCES:
- [Derived] Thierry S, Jaulin F, Starck C, Aries P, Schmitz J, Kerkhoff S, Bernard CI, Komorowski M, Warnecke T, Hinkelbein J. Evaluation of free-floating tracheal intubation in weightlessness via ice-pick position with a direct laryngoscopy and classic approach with indirect videolaryngoscopy. NPJ Microgravity. 2023 Sep 8;9(1):73. doi: 10.1038/s41526-023-00314-y. PMID 37684267